CLINICAL TRIAL: NCT03402919
Title: The Comprehensive Assessment of Neurodegeneration and Dementia Study
Brief Title: Comprehensive Assessment of Neurodegeneration and Dementia
Acronym: COMPASS-ND
Status: Recruiting | Type: Observational
Sponsor: McGill University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alzheimer Society of Canada (Other); Sanofi (Industry); New Brunswick Health Research Foundation (Other); Saskatchewan Health Research Foundation (Other); Michael Smith Foundation for Health Research (Other); Nova Scotia Health Research Foundation (Other Government); Eli Lilly and Company (Industry); Canadian Nurses Foundation (CNF) (Other); Ontario Brain Institute (Other); Pfizer (Industry); Canadian Consortium on Neurodegeneration in Aging (Other)
Responsible Party: Principal Investigator, Howard Chertkow, Principal Investigator, Baycrest
Other Study IDs: CCNA 2015
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Dementia; Mild Cognitive Impairment (MCI); Subjective Cognitive Impairment; Parkinson's Disease (PD); Lewy Body Disease(LBD); Mixed Dementia; Frontotemporal Dementia (FTD); Alzheimer Disease (AD); Cognitively Unimpaired; Subjective Cognitive Decline (SCD)
Keywords: Observational; Dementia; Alzheimer's Disease; Parkinson's Disease; Biosample; Genetics; Neuropsychological; MRI; Microbiome; Plasma
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Parkinson Disease; Lewy Body Disease; Mixed Dementias; Frontotemporal Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Saliva, Urine, Fecal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Normal healthy elderly: participants with no subjective or objective cognitive deficits or decline.
- Subjective Cognitive Decline: Participants with a complaint of subjective cognitive impairment, but no objective evidence of such.
- Mild Cognitive Impairment (MCI): Participants with objective evidence of cognitive impairment, but it does not impact on daily function.
- Vascular MCI: Participants meeting criteria of MCI who also show signs of cerebrovascular disease on imaging but have no history of stroke.
- Alzheimer's Disease: Participants with dementia of the Alzheimer's type according to the National Institute of Aging-Alzheimer's Association criteria
- Dementia of Mixed Etiology: Participants with dementia and evidence of more than one etiology.
- Lewy Body/Parkinson's spectrum: Participants with Parkinson's disease who show mild or moderate cognitive impairment and/or dementia.
- Frontotemporal dementia (FTD) spectrum: Participants with behavioral variant FTD, primary progressive aphasia, progressive supranuclear palsy, or corticobasal syndrome

SUMMARY:
This is a longitudinal observational study recruiting individuals between the ages of 50 and 90 with different types of dementia as well as a comparison group without cognitive deficits. Participants are/will be recruited at sites across Canada and will undergo assessments, neuroimaging, and biological sample collection.

DETAILED DESCRIPTION:
This is a longitudinal observational study that started in Phase I with the recruitment of 1173 participants between the ages of 50 and 90 years with Subjective Cognitive Impairment, Mild Cognitive Impairment, Mild Cognitive Impairment with subcortical vascular lesions, Alzheimer's Disease, Mixed dementia, Lewy Body Dementia, Parkinson's Disease Dementia, Parkinson's Disease with Mild Cognitive Impairment and Frontotemporal Dementia as well as healthy elderly subjects without cognitive complaints or deficits. These participants were enrolled in 30 different centres across Canada.

All subjects involved in the study underwent rigorous evaluations at baseline, including clinical assessment, neuropsychological assessment, genomics and neuroimaging. Biological samples from blood, saliva, urine, fecal matter, buccal cells and cerebrospinal fluid were collected, stored, and analyzed.

Longitudinal follow-up determining if there has been any change in their diagnosis was carried out annually and longitudinal re-evaluation was carried out at two times: Time 2 and Time 3.

In Time 3, 400 participants across the non-dementia cohorts (Cognitively Unimpaired, Subjective Cognitive Impairment, Mild Cognitive Impairment, Mild Cognitive Impairment with a Vascular Component, Parkinson's Disease with no Cognitive Impairment, Parkinson's Disease with Mild Cognitive Impairment) with up to 12 years of education will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Has subjective or objective cognitive impairment
* Written informed consent must be obtained and documented (from the patient or, where jurisdictions allow it, from a caregiver/family member)
* Sufficient proficiency in English or French to undertake self report and neuropsychological testing
* Geographic accessibility to the study site
* Must have a study partner who can participate as required in the protocol (provide corroborative information)
* Up to 12 years of education
* Fits into one of the following groups: Cognitively Unimpaired, Subjective Cognitive Impairment, Mild Cognitive Impairment, Vascular Mild Cognitive Impairment, Parkinson's Disease, Parkinson's Disease with Mild Cognitive Impairment

Exclusion Criteria:

* The presence of other significant known chronic brain disease such as: moderate to severe chronic static leukoencephalopathy (including previous traumatic injury), multiple sclerosis, a serious developmental handicap, malignant tumors, Parkinson's disease (other than for the Parkinson's cohort), and other rarer brain illnesses
* Ongoing alcohol or drug abuse which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures
* Symptomatic stroke within the previous year
* Unable to undergo MRI scan due to medical contraindications or inability to tolerate the procedure

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2300 English and/or French-speaking participants recruited from across Canada in the following groups:
  * 650 Cognitively healthy volunteers
  * 300 volunteers with Subjective Cognitive Decline
  * 400 volunteers with Mild Cognitive Impairment
  * 200 volunteers with Vascular Mild Cognitive Impairment
  * 150 volunteers with Alzheimer's disease
  * 200 volunteers with Dementia of Mixed Etiology
  * 200 volunteers with Parkinson's disease and cognitive impairment
  * 200 volunteers with Frontotemporal spectrum dementia
Sampling Method: Non-Probability Sample
Enrollment: 1573 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) score | 8 years
  change in MoCA total score. The MoCA is a test of global cognition scored out of 30 with a higher score indicating better performance. The minimum score is 0 and the maximum score is 30.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borrie, MD, Study Director — Western University; Natalie Philips, PhD, Study Director — Concordia University, Montreal; Jaspreet Bhangu, MB, Study Director — Western University
Locations (19):
- Canada (19):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Djavad Mowafaghian Centre for Brain Health, Vancouver, British Columbia
  - Island Health, Victoria, British Columbia
  - Veteran's Memorial Building, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Health Care London, London, Ontario
  - Gait and Brain Lab, London, Ontario
  - Bruyère Research Institute, Ottawa, Ontario
  - Kawartha Centre, Peterborough, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network Memory Clinic, Toronto, Ontario
  - Baycrest Clinical Unit, Toronto, Ontario
  - University of Waterloo, Waterloo, Ontario
  - Research Institute of the McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital/McGill Memory Clinic, Montreal, Quebec
  - Clinique de cognition Institut universitaire de gériatrie de Montréal, Montreal, Quebec
  - Hôpital Enfant-Jésus, Québec, Quebec
  - Centre de recherche sur le vieillissement CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared initially with all Canadian Consortium on Neurodegeneration and Aging (CCNA) affiliated researchers and eventually with all interested researchers internationally.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data is currently available.
Access Criteria: Reaserchers who which to access the database will be required to create an account through CCNA and demonstrate their research credentials and their affiliation to a recognized research organization. Users must confirm that their intended use of data respects CCNA policies and applicable ethical, legal, and data governance requirements. Researchers are further required to hold data secure, not to attempt the re-identification of research participants, and not to perform research that could cause communities to experience stigmatization or discrimination.
URL: https://ccna-ccnv.ca/wp-content/uploads/2025/07/Data-Access-and-Data-Query-Tool-MANUAL-OF-PROCEDURES-v3.1-July-2025.pdf

REFERENCES:
- [Derived] Montero-Odasso M, Sarquis-Adamson Y, Kamkar N, Pieruccini-Faria F, Bray N, Cullen S, Mahon J, Titus J, Camicioli R, Borrie MJ, Bherer L, Speechley M. Dual-task gait speed assessments with an electronic walkway and a stopwatch in older adults. A reliability study. Exp Gerontol. 2020 Dec;142:111102. doi: 10.1016/j.exger.2020.111102. Epub 2020 Oct 2. PMID 33017671
- See also: This is a direct link to the study's website. — https://ccna-ccnv.ca/compass-nd-study/
- See also: CIHR COMPASS-ND Study — https://cihr-irsc.gc.ca/e/53979.html

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03402919/Prot_SAP_000.pdf
  • Informed Consent Form: Study Participant Informed Consent Form (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03402919/ICF_001.pdf
  • Informed Consent Form: Study Partner Informed Consent Form (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03402919/ICF_002.pdf